CLINICAL TRIAL: NCT06460012
Title: Support Via Technology: Living and Learning With Advancing Dementia-REVISED
Acronym: STELLA-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Hart Family Foundation (Unknown)
Responsible Party: Principal Investigator, Allison Lindauer, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00025741
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Caregiver Burden
Keywords: caregivers; dementia; RMBPC; caregiver support
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: Care partners will participate in a self-directed, 8-week online course via the STELLA-R website, followed by 8-weeks of unrestricted access to the website, with 8 weeks of restricted access. One group will receive the 8-week online course followed by the 8-week unrestricted access immediately after enrolling. The other group will receive the 8-week online course and 8-week unrestricted access 2 months after enrolling.
Who Masked: Participant
Masking Description: Care partners will be randomized into one of two groups. Care partners will be blinded to which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Care partners start the STELLA-R Curriculum immediately after enrollment.
  Interventions: Behavioral: STELLA-R Curriculum; Behavioral: Unrestricted Access; Behavioral: Limited Access
- Waitlist Control Group (Active Comparator): Care partners start the STELLA-R Curriculum 8 weeks after enrollment.
  Interventions: Behavioral: STELLA-R Curriculum; Behavioral: Unrestricted Access; Behavioral: Limited Access

INTERVENTIONS:
Behavioral: STELLA-R Curriculum — The STELLA-R curriculum is presented utilizing the ABC analytic approach to address care recipient's distressing behaviors. Using the scaffold of the ABC pyramid, they will receive video instructions on how to fully define the Behaviors they want to address by observing, describing, and writing about them. The care partners will learn to identify the Activators, the triggers for the behaviors. Next, care partners will learn to consider what happens after the behaviors, the Consequences. This is an 8-week self-directed, online weekly curriculum.
Behavioral: Unrestricted Access — Following the STELLA-R curriculum, care partners will receive 8 weeks of unrestricted access to all lessons and resources.
  Other Names: Post-Intervention Phase; Review Phase
Behavioral: Limited Access — Experimental and Waitlist Control group will experience 8 consecutive weeks of limited access to the STELLA-R website and resources. Waitlist Control will experience this from Week 1 to Week 8 while the Experimental Group will reach this phase from Week 17 to Week 24.
  Other Names: Restricted Access

SUMMARY:
STELLA-R is a multicomponent, self-directed, online intervention designed to facilitate effective management of behavioral and psychological symptoms that are common in many types of dementia. The curriculum instructs care partners to use the ABC approach, a cognitive behavioral technique that teaches care partners to describe a Behavior, then consider the Activators and Consequences of a care recipient behavior. The goal of this intervention is to reduce care partner burden and decrease reactivity to upsetting behaviors.

DETAILED DESCRIPTION:
Providing care for a family member with Alzheimer's disease and related dementias (ADRD, aka, "dementia") is both rewarding and risky. Care partners exposed to chronic stress, often over years, are susceptible to physical and psychological ailments. Dementia involves neurodegeneration and those affected typically depend on family members for support and physical care. The "care partners" for those with dementia often experience concerning psychological and physical outcomes due to the demands of caregiving. No matter what type of dementia, most care partners experience some burden. The burden is often related to the behavioral symptoms that most people with dementia experience.

Care partners for those with dementia experience burden, grief, exhaustion and physical ailments. Programs for these care partners are more available. Effective interventions that reduce care partner burden and health risks are also available, but various factors impede participation, including distance, cost, behavioral symptoms of dementia, stigma and social anxiety. Recognizing the need to reduce barriers to access, scientists have turned to internet-based interventions.

The STELLA suite of research studies addresses the need for easily accessible, effective interventions designed to reduce burden in care partners for those with dementia. These studies examine the acceptability, feasibility, and efficacy of interventions modeled on Teri's psychoeducational behavior change intervention. We have completed two pilot studies for care partners for those with dementia using interventions with the STELLA-R precursor. These studies found early efficacy and acceptability for the intervention. We are currently testing a STELLA intervention which uses objective, technology-based assessments (OHSU IRB # 19306) and another, larger study which tests a STELLA intervention with a large national sample (OHSU IRB # 22288; NIA R01AG067546). In addition, with funding from the Association for Frontotemporal Degeneration (AFTD) we tested a similar intervention (STELLA-FTD) for care partners caring for a family member with frontotemporal dementia (OHSU IRB # 22721).

In all STELLA studies care partners work with professional guides to use the ABC analytic approach to describe a distressing behavior, then identify its activators and consequences. With this information, care partners can develop plans to reduce behavioral symptoms. In this proposed study, we will assess an online version of Tele-STELLA.

STELLA-R is informed by the World Health Organization (WHO) guidance to include rehabilitation science in dementia care to facilitate effective management of the advancing behavioral, communication, physical and social changes that come with progressive neurodegenerative dementias (e.g., Alzheimer's disease, frontotemporal degeneration, Lewy Body dementia). Grounded in self-efficacy theory and foundational research, STELLA-R will train care partners to address current behavioral symptoms and prepare for future ones.

The specific aims of this study are:

Aim 1. Assess feasibility and acceptability of STELLA-R

Aim 2. Compare the efficacy of STELLA-R in reducing care partner reactivity to dementia-related behavioral symptoms between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult caring for family member with ADRD
* Age of 18 years or older
* Speaks and understands English to be able to participate in intervention
* Owns a telephone (smartphone, cell phone or landline)
* Has email and mailing address to receive study materials and surveys
* Provides informed consent to participate in the research
* Lives in Oregon, Washington or Idaho
* Identifies two or more behavioral symptoms that are distressing to them (care partner)

Exclusion Criteria:

* Vision problems severe enough to prevent participation
* Unwilling or unable to adequately follow study instructions and participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Revised Memory and Behavior Problems Checklist (RMBPC) | Week 1, Week 8, Week 16, Week 24
  The primary outcome variable, reactivity, will be assessed with the RMBPC, which measures the frequency of care recipient behavioral symptoms and care partner reactions to these behaviors. The RMBPC was chosen because it aligns with our theoretical foundation that assumes burden is a result of care partner reactions to behavioral symptoms.
  The RMBPC is a 29-item caregiver report measure, 5-point Likert scale with frequency measuring from 0 (never occurred) to 4 (daily or more often) and reactivity measuring from 0 (not at all) to 4 (extremely) for a total score between 0-116 for each subscale (frequency subscale and reactivity subscale). Higher scores indicate greater behavioral problems.
Feasibility of STELLA-R Intervention | 10 months
  We will assess the feasibility of implementing STELLA-R across Oregon, Washington and Idaho. We will analyze metadata from the STELLA-R website to assess care partner usage of intervention materials. We will assess data from the surveys to characterize the sample, assess program acceptability, and measure treatment fidelity. We will compare demographic information, computer use, health-care usage, behavioral symptom frequency, medication use, care partner reactivity, burden and depression.
Acceptability of STELLA-R Intervention | Week 24
  For acceptability, we will utilize the STELLA-R Experience Survey which is a 16-item survey on satisfaction, privacy, and ease of use. We will analyze the STELLA-R Experience Survey results using descriptive statistics. We will identify themes of acceptance, or lack thereof, of STELLA-R and the underpinnings of their impressions.

SECONDARY OUTCOMES:
Fortinsky's Measurement of Family Care Partner Self-Efficacy for Managing Dementia | Week 1, Week 8, Week 16, Week 24
  Self-efficacy, the mediating variable, will be assessed using Fortinsky's measurement of family care partner self-efficacy for managing dementia. Fortinsky's assess the targets in STELLA-R: behavior symptom management and service use.
  Fortinsky's measurement is a 9-item Likert scale ranging from 1 (not at all certain) to 10 (very certain). Higher scores are associated with fewer depressive symptoms and fewer physical health symptoms.
Preparedness for Caregiving Scale | Week 1, Week 8, Week 16, Week 24
  The Preparedness for Caregiving Scale is a 10-item Likert scale ranging from 0 (not at all prepared) to 4 (very well prepared). We will measure care partner preparedness for current and future challenges to test the effect of a group-based intervention.
Ten-Item Personality Inventory (TIPI) | Week 1
  The Ten-Item Personality Inventory is a 10-item Likert scale measure to assess introversion and extraversion. Choices range from 1 (disagree strongly) to 7 (agree strongly) with reverse scoring on items 2, 4, 6, 8 and 10. Scoring on items are as follows: extraversion: 1, 6R; agreeableness: 2R, 7; conscientiousness: 3, 8R; emotional stability: 4R, 9; openness to experiences: 5, 10R. We will use this measure to test the effect of a group-based intervention.
Personalized Target Behavior Survey | Week 1, Week 8
  The Personalized Target Behavior Survey measure frequency and reactivity of up to 3 personalized behaviors identified by care partners. We will collect data on the number of ABC plans each care partner writes on the Orbit weekly survey and the STELLA-R website.
Emotional and Physical Strain | Weekly for 6 months
  The Orbit weekly survey will measure emotional and physical strain for caregivers.
Healthcare Use | Weekly for 6 months
  The Orbit weekly survey will measure service use and medication use for behavioral symptoms.
Zarit Burden Interview | Weekly for 6 months
  The Orbit weekly survey will include the Zarit Burden Interview, a 4-item caregiver report measuring care partner burden. This measure is a 5-point Likert scale with a range of 0 (never) to 4 (nearly always) with higher scores meaning greater burden.
The Neuropsychiatric Inventory (NPI-Q) | Week 1, Week 8, Week 16, Week 24
  The NPI-Q with Caregiver Self-Efficacy Scale evaluates 12 behavioral disturbances in dementia. Each domain captures severity of BPSD and caregiver self-efficacy. Severity is rated 1 (mild) to 3 (severe) and self-efficacy is reverse scored from 4 (not at all confident) to 1 (very confident). This measure assesses self-efficacy in addressing specific behavioral symptoms.
Placement Plan Scale | Week 1, Week 8, Week 16, Week 24
  1-item Likert scale assessment of plans for placement of family member with dementia. Care partners will rate their likelihood of moving their family member with dementia to another living arrangement from 1 (not at all likely) to 5 (very likely).
Use of Professional Services | Week 1, Week 8, Week 16, Week 24
  A 7-item binary assessment of professional services used to address their family member with dementia's needs in the past 2 months. Care partners will answer Yes or No to using a: dietitian, elder care attorney, occupational therapist, physical therapist, psychologist, social worker, speech therapist, and healthcare professional.
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Week 1, Week 24
  A 12-item assessment measuring mindfulness, distress, well-being, emotion-regulation, and problem-solving approaches. A Likert scale ranging from 1 (rarely/not at all) to 4 (almost always) with reverse scoring on items 2, 6 and 7.
Pittsburgh Sleep Quality Index (PSQI) | Week 1, Week 24
  The PSQI contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available) that assesses self-rated sleep quality and disturbances over a 1-month time interval. Only self-rated questions are included in scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. A score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points. "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
ABC Plans | Week 8, Week 16, Week 24
  A 1-item measure to assess total quantity of ABC plans created. Options are 1 (1-3), 2 (4-6), 3 (7-9) or 4 (10 or more). Experimental group completes this measure on weeks 8, 16 and 24. Wait-list control group completes this measure on weeks 16 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lindauer, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Layton Aging and Alzheimer's Disease Research Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon request to our Alzheimer's Disease Research Center.
Supporting Information: Study Protocol
Time Frame: Once data is available, it will be available indefinitely.
Access Criteria: Requests need to be made to the PI at the Oregon Alzheimer's Disease Research Center (OARDC). A short data request form will need to be submitted.